CLINICAL TRIAL: NCT03344198
Title: Effects of Combined Diet & Exercise Intervention on Cardiovascular Risk Factors in Firefighters & Civilians
Brief Title: Exercise & Diet Effects on CV Risk in Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Hampshire (Other)
Collaborators: American Heart Association (Other); California State University, San Marcos (Other)
Responsible Party: Principal Investigator, Deborah Feairheller, Assistant Professor, California State University, San Marcos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 005-8242-01
Record Dates: First submitted 2017-10-24; First posted 2017-11-17 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Risk Factor; Blood Pressure; Exercise; Diet Modification; Health Promotion
Keywords: Cardiovascular Disease; Mediterranean Diet; Exercise Training; Blood Pressure
MeSH Terms: conditions — Motor Activity; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Firefighter (Veteran) Group (Experimental): Firefighters with >10yrs experience. Circuit Training exercise & Modified Mediterranean diet
  Interventions: Behavioral: Circuit Training exercise & Modified Mediterranean diet
- Firefighter (Novice) Group (Experimental): Firefighters with <10yrs experience. Circuit Training exercise & Modified Mediterranean diet
  Interventions: Behavioral: Circuit Training exercise & Modified Mediterranean diet
- Control Non-Firefighter Group (Experimental): Non-Firefighter adults. Circuit Training exercise & Modified Mediterranean diet
  Interventions: Behavioral: Circuit Training exercise & Modified Mediterranean diet

INTERVENTIONS:
Behavioral: Circuit Training exercise & Modified Mediterranean diet — Participants will receive circuit training program and a modified Mediterranean diet program. Educational sessions, serving size training, and portion containers will be provided. Participants will also receive individualized support throughout the 6 week intervention.

SUMMARY:
The study will explore the capacity for a lifestyle modification in firefighters to improve blood pressure, blood vessel stiffness, inflammation, and reduce oxidative stress. The study will be a pre- post-testing controlled trial with three groups. The intervention will be a weekly circuit workout program and a Mediterranean (high fruit/vegetable) diet. The groups will be firefighters with >10yrs experience, firefighters with <10yrs experience, and control Non-firefighters.

DETAILED DESCRIPTION:
Recent statistics from the American Heart Association (AHA) have reported that >92% of adults in the U.S. meet at least 1 metric for cardiovascular disease risk factors. In firefighters, this increased risk is especially concerning. The National Fire Protection Agency (NFPA) estimates there are around 1.3 million firefighters in the United States, 70% of which are volunteer. The prevalence of impaired cardiovascular health is higher in firefighters than in the general population and the leading line-of-duty death (LODD) cause is cardiac related. It is known that exercise and diet mitigate cardiovascular disease risk. Meeting the physical activity guidelines remains a target of ideal cardiovascular health and a major public health concern. However, the NFPA does not require volunteer fire companies to have a fitness program for their crew, and sadly less than a third of the stations actually do. And importantly, cardiovascular-related LODD remains a major issue in the firefighter population. The results could guide clinical treatment for firefighters and may therefore reduce cardiac-related LODD.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Able to Exercise

Exclusion Criteria:

* More than one anti-hypertensive medication
* More than one cholesterol medication
* Diabetic
* Prior Cardiac incident

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Pre-Intervention (Week 0), Post-Intervention (Week 6)
  Blood pressure surge response to alarm will be measured by ambulatory blood pressure monitor

SECONDARY OUTCOMES:
Change in vascular stiffness | Pre-Intervention (Week 0), Post-Intervention (Week 6)
  Stiffness will be measured by pulse wave velocity
Change in cardiopulmonary fitness | Pre-Intervention (Week 0), Post-Intervention (Week 6)
  Fitness will be measured by treadmill test
Change in body composition | Pre-Intervention (Week 0), Post-Intervention (Week 6)
  Body composition will be measured by bioelectrical impedance
Change in inflammation | Pre-Intervention (Week 0), Post-Intervention (Week 6)
  Inflammation will be measured by assay of circulating bio-markers through blood draw.
Change in oxidative stress | Pre-Intervention (Week 0), Post-Intervention (Week 6)
  Oxidative stress will be measured by assay of circulating antioxidant bio-markers through blood draw.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L Feairheller, PhD, Principal Investigator — California State University, San Marcos
Locations (1):
- California State University San Marcos, San Marcos, California, United States

IPD SHARING:
Plan to Share IPD: Yes
data will be entered
Supporting Information: Analytic Code
Time Frame: 2023
Access Criteria: must get approval from PI

REFERENCES:
- [Background] Donahue S, McMorrow C, Almeida AA, Feairheller DL. Feasibility and Perception of a Diet and Exercise Intervention Delivered via Telehealth to Firefighters. Int J Telerehabil. 2022 Jun 3;14(1):e6458. doi: 10.5195/ijt.2022.6458. eCollection 2022. PMID 35734390
- [Background] Almeida AA, Reeve EH, Dickinson RL, Carty M, Gilpin J, Feairheller DL. Civilians Have Higher Adherence and More Improvements in Health With a Mediterranean Diet and Circuit Training Program Compared With Firefighters. J Occup Environ Med. 2022 Jun 1;64(6):488-494. doi: 10.1097/JOM.0000000000002478. Epub 2022 Jan 4. PMID 34985026
- [Background] Feairheller DL, Smith M, Carty M, Reeve EH. Blood pressure surge with alarm is reduced after exercise and diet intervention in firefighters. Blood Press Monit. 2023 Jun 1;28(3):134-143. doi: 10.1097/MBP.0000000000000649. Epub 2023 Apr 12. PMID 37070561
- [Background] McLaughlin KC, Perez AN, Donahue S, Feairheller DL. Tactical Circuit Training Improves Blood Pressure and Vascular Health More Than Resistance Training. Int J Exerc Sci. 2021 Nov 1;14(3):1320-1333. doi: 10.70252/CKXH1603. eCollection 2021. PMID 35096239
- [Background] Rynne PJ, Derella CC, McMorrow C, Dickinson RL, Donahue S, Almeida AA, Carty M, Feairheller DL. Blood pressure responses are dependent on call type and related to hypertension status in firefighters. Blood Press. 2023 Dec;32(1):2161997. doi: 10.1080/08037051.2022.2161997. PMID 36597210
- [Background] McMorrow C, Feairheller DL. Blood Pressure Responses in Firefighters: A Review. Curr Hypertens Rev. 2022;18(2):145-152. doi: 10.2174/1573402118666220103094201. PMID 34979891
- [Background] Derella CC, Aichele KR, Oakman JE, Cromwell CM, Hill JA, Chavis LN, Perez AN, Getty AK, Wisdo TR, Feairheller DL. Heart Rate and Blood Pressure Responses to Gear Weight Under a Controlled Workload. J Occup Environ Med. 2017 Apr;59(4):e20-e23. doi: 10.1097/JOM.0000000000000997. PMID 28628053

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT03344198/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT03344198/ICF_001.pdf